CLINICAL TRIAL: NCT02666794
Title: Plasmatic Catecholamines After Neuraxial Labor Analgesia: a Randomized Controlled Trial Comparing Epidural Versus Combined Spinal-epidural
Brief Title: Plasmatic Catecholamines: Randomized Controlled Trial Comparing Epidural Versus Combined Spinal-epidural
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, SHIRLEY ANDRADE SANTOS, Anesthesiologist, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 45992815000000068
Record Dates: First submitted 2015-12-21; First posted 2016-01-28 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Fetal Bradycardia; Hypertonic Uterine; Catecholamines
Keywords: analgesia; fetal bradycardia; hypertonic uterine
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puncture epidural (Active Comparator): Women in labor the epidural group will receive epidural bupivacaine with vasoconstrictor 0.125% 10 ml plus 20 micrograms sufentanil, followed by the placement of the epidural catheter
  Interventions: Drug: Epidural bupivacaine with vasoconstrictor 0.125%; Drug: Epidural sufentanil; Procedure: Placement of the epidural catheter
- Puncture combined spinal-epidural (Active Comparator): The mothers of the combined spinal-epidural analgesia group will receive intrathecal hyperbaric bupivacaine solution 0.5% 2.5 mg plus 5.0 micrograms of sufentanil and plus 60 micrograms of morphine, followed by placement of an epidural catheter to the catheter through technical needle
  Interventions: Drug: Intrathecal hyperbaric bupivacaine solution 0.5%; Drug: Intrathecal morphine; Procedure: Placement of an epidural catheter to the catheter through technical needle; Drug: Intrathecal sufentanil

INTERVENTIONS:
Drug: Epidural bupivacaine with vasoconstrictor 0.125% — 10 ml
  Arms: Puncture epidural
Drug: Epidural sufentanil — 20 mcg
  Arms: Puncture epidural
Procedure: Placement of the epidural catheter — Placement of the epidural catheter
  Arms: Puncture epidural
Drug: Intrathecal hyperbaric bupivacaine solution 0.5% — 2.5 mg
  Arms: Puncture combined spinal-epidural
Drug: Intrathecal morphine — 60 mcg
  Arms: Puncture combined spinal-epidural
Procedure: Placement of an epidural catheter to the catheter through technical needle — Placement of an epidural catheter to the catheter through technical needle
  Arms: Puncture combined spinal-epidural
Drug: Intrathecal sufentanil — 5 mcg
  Arms: Puncture combined spinal-epidural

SUMMARY:
Combined spinal-epidural (CSE) for labor analgesia has been associated with fetal bradycardia and uterine hypertonia, possibly due to asymmetric decrease in catecholamine levels, when compared with epidural analgesia (EP).

DETAILED DESCRIPTION:
Background: Combined spinal-epidural technique for labor analgesia has been associated with fetal bradycardia and uterine hypertonia, when compared with epidural analgesia, possibly due to asymmetric decrease in catecholamine levels (epinephrine and norepinephrine) following neuraxial block. However, there are no studies comparing plasmatic catecholamine levels between those two techniques. This study aimed to compare spinal-epidural versus epidural regarding pre and post-analgesia catecholamine levels, uterine tone and fetal heart rate.

Methods: Randomized clinical trial with 47 laboring patients divided in two groups. Primary outcome was plasmatic catecholamine measurements before and after neuraxial block. Secondary outcomes were fetal heart rate changes, uterine hypertonia, hypotension episodes, pain relief and fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

Parturients aged over 18 years were included when they requested labor analgesia. The inclusion criteria were: patients between 37 and 42 gestational weeks, single pregnancy, in active labor (induced or spontaneous), requesting analgesia with 7 cm or less of cervical dilation. As it is a center that attends only high-risk pregnancies, ASA II or III

Exclusion Criteria:

Contraindications to interventions, either due to severe comorbidity or contraindication to neuraxial block; previous use of systemic opioids during labor, maternal amniotic infection or known fetal diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Cathecolamines levels | at the moment of analgesia and 20 minutes after
  Pattern of cathecolamines levels
Fetal bradycardia | 15 minutes before analgesia and 30 minutes after continuously
  Fetal bradycardia is defined as the baseline drops to less than 100 bpm
Increase in uterine tone | 15 minutes before analgesia and 30 minutes after continuously
  Increase in uterine tone (qualitative measure)

SECONDARY OUTCOMES:
Maternal hipotension | 30 minutes after analgesia (measures every 5 minutes)

OTHER OUTCOMES:
Pain scores | 20 minutes after analgesia (measures every 5 minutes)
APGAR score | At birth
Fetal acidosis | At birth
  umbilical arterial blood

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Santos, MD, Principal Investigator — Anesthesiologist
Locations (1):
- Shirley Andrade Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baschat AA. Fetal growth restriction - from observation to intervention. J Perinat Med. 2010 May;38(3):239-46. doi: 10.1515/jpm.2010.041. PMID 20205623
- [Result] Abrao KC, Francisco RPV, Miyadahira S, Cicarelli DD, Zugaib M. Elevation of uterine basal tone and fetal heart rate abnormalities after labor analgesia: a randomized controlled trial. Obstet Gynecol. 2009 Jan;113(1):41-47. doi: 10.1097/AOG.0b013e31818f5eb6. PMID 19104358
- [Result] Van de Velde M, Vercauteren M, Vandermeersch E. Fetal heart rate abnormalities after regional analgesia for labor pain: the effect of intrathecal opioids. Reg Anesth Pain Med. 2001 May-Jun;26(3):257-62. doi: 10.1053/rapm.2001.22258. PMID 11359226
- [Result] Nielsen PE, Erickson JR, Abouleish EI, Perriatt S, Sheppard C. Fetal heart rate changes after intrathecal sufentanil or epidural bupivacaine for labor analgesia: incidence and clinical significance. Anesth Analg. 1996 Oct;83(4):742-6. doi: 10.1097/00000539-199610000-00014. PMID 8831313
- [Result] Collis RE, Davies DW, Aveling W. Randomised comparison of combined spinal-epidural and standard epidural analgesia in labour. Lancet. 1995 Jun 3;345(8962):1413-6. doi: 10.1016/s0140-6736(95)92602-x. PMID 7760614
- [Result] Nakamura G, Ganem EM, Rugolo LM, Castiglia YM. Effects on mother and fetus of epidural and combined spinal-epidural techniques for labor analgesia. Rev Assoc Med Bras (1992). 2009 Jul-Aug;55(4):405-9. doi: 10.1590/s0104-42302009000400014. PMID 19750306
- [Result] Patel NP, El-Wahab N, Fernando R, Wilson S, Robson SC, Columb MO, Lyons GR. Fetal effects of combined spinal-epidural vs epidural labour analgesia: a prospective, randomised double-blind study. Anaesthesia. 2014 May;69(5):458-67. doi: 10.1111/anae.12602. PMID 24738803
- [Result] Simmons SW, Taghizadeh N, Dennis AT, Hughes D, Cyna AM. Combined spinal-epidural versus epidural analgesia in labour. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD003401. doi: 10.1002/14651858.CD003401.pub3. PMID 23076897